CLINICAL TRIAL: NCT03057223
Title: Three-Dimensional Printing of Patient-Specific Titanium Plates in Jaw Surgery: An Open-Label, Prospective Pilot Clinical Study
Brief Title: Three-Dimensional Printing of Patient-Specific Titanium Plates in Jaw Surgery: A Pilot Study
Acronym: 3DJP16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yuxiong Su, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: UW 16-315
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Mandibular Neoplasms; Maxillary Neoplasms; Dentofacial Deformities; Maxillofacial Injuries
Keywords: 3D printing; patient-specific titanium plate; mandibular malignancy; dento-maxillofacial deformity; orthognathic surgery; mandibular reconstruction
MeSH Terms: conditions — Mandibular Neoplasms; Maxillary Neoplasms; Dentofacial Deformities; Maxillofacial Injuries

STUDY DESIGN:
Intervention Model Description: This is an open-label, prospective, single-arm, and single-center interventional clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3D Jaw Plate (Experimental): 3D Jaw Plate will be used in internal fixation.
  Interventions: Device: 3D-printed patient-specific titanium plates

INTERVENTIONS:
Device: 3D-printed patient-specific titanium plates — 3D-printed patient-specific titanium plates will be used in patients.
  Other Names: 3D Jaw Plate

SUMMARY:
Medical titanium plates are routinely used in fixing mobilized bone segments in jaw surgeries. Generally these plates are commercialized with standard construction specifications. Thus they should be repeatedly bended and arched to match the contour of anchored jaw bones before located in place and fastened by screws. To prevent stress fatigue induced by plate bending and improve structural design, we utilized the three-dimensional printing technique and developed a new production procedure in fabricating customized titanium plates according to each patient's specific skeletal contours and dimensions derived from medical imaging data. In general, the three-dimensional printing of customized implants are expected to facilitate surgical operation, reduce application duration and improve precise restoration.

Up until now, the application of three-dimensional printing of titanium fixation plates in jaw surgery has been available only at two centers globally. The published preliminary work have proved the prospect of customized titanium plates in promoting mandibular reconstruction surgery and upper maxilla orthognathic surgery though their printed titanium plates looked rather bulky and the sample sizes were small and there is still lack of qualified randomized controlled trials between the printed and the conventional titanium plates. To better benefit from the burgeoning use of three-dimensional printing in health care, it is imperative to conduct a feasibility study in exploring the application of three-dimensional printing of titanium fixation plates in jaw surgery based on our patients.

The aim of the study is to conduct a case series study focusing on the feasibility and safety of applying three-dimensional printed titanium plates in jaw reconstruction surgery and orthognathic surgery. The outcome measures include the success rate, potential adverse events and accuracy. A sample size of 48 subjects will be recruited prospectively. Considering the facts that titanium plates are widely used in jaw surgery and our unit is the largest oral and maxillofacial surgery center in Hong Kong, the well-designed customized titanium plate is therefore with great potential benefit for the patients in our population. Furthermore, the well-developed three-dimensional manufacturing protocol could also be applied in other relevant medical areas and push forward the personalized medicine era in the future.

DETAILED DESCRIPTION:
Plate osteosynthesis is the basic philosophy in maintaining skeletal stabilization in jaw surgery. Numerous branded osteosynthesis systems are available and most of them are made from pure titanium or titanium alloys with standard construction specifications. Usually these titanium plates should be bended and arched to better match the three-dimensional contour of anchored jaw bones. However the optimal bending of the titanium plate sometimes is difficult and time-consuming especially for the inexperienced surgeons and in complicated cases. Excessive bending could also initiate residual stress and potentially worsen the mechanical properties of titanium plates(1).

The three-dimensional (3D) printing, or additive manufacturing, has been well developed in fabricating customized materials from the computer-generated digital files. In recent years, 3D printing of patient-specific medical implants has been evolving with the newly-emerged technology of powder bed fusion, which enabled the melting of metals and further shaping of devices(2). In September 2015, China's innovative 3D printed hip joint prosthesis was commercially certified by China's State Food and Drug Administration. In February 2016, the world's first 3D printed patient-specific titanium cranial/craniofacial plate implant got the U.S. Food and Drug Administration's approval. Beyond that, a number of other printed implants have showed excellent performance in clinical research. These printed medical implants are majorly from pure titanium or Ti6Al4V alloy, which exhibit good resistance to fatigue and corrosion and are considered the most biocompatible metal(3). Relying on individualized imaging data, the printed implants are patient-specific and adapt to the anatomical structures precisely. Since the additive manufacturing is ultimately different from the conventional multi-step production operations, it could reduce costs and lead times, especially in printing complex devices for individualized cases. While in clinical applications, 3D printing of customized implants are expected to facilitate surgical operation, reduce application duration and improve precise restoration(4). It is predicted the application of 3D printing technique in medical area may bring forward another major advance toward personalized medicine(5). Many more customized medical implants will be approved in the future across the world.

With the advent of metal additive manufacturing, the 3D-printed patient-specific titanium plates have been successfully fabricated. In 2012, Per Derand et al. reported the first application of 3D-printed titanium plates with the established workflow from imaging, via virtual design, to manufacturing of cutting guide and customized titanium reconstruction plates, and its utility in the fibula-based mandibular reconstruction surgery. The pre-printed plates did facilitate the operation and reduced the operation duration about half an hour though the postoperative accuracy of the grafted bone was modest compared with the virtual planning(6). Simultaneously, Leonardo Ciocca et al. reported the computer-aided designing and manufacturing in guiding secondary mandibular reconstruction of a discontinuity defect involving the employment of the surgical guide and printed titanium reconstruction plate in surgical transferring of virtual planning(7). In 2013, Simona Mazzoni and Leonardo Ciocca et al. applied the same surgical protocol in a study group of seven mandibular reconstruction patients and compared its advantages with the standard pre-plating technique on stereolithographic models in a control group. The results revealed the computer-aided surgical protocol was viable in reproducing the patients' anatomical contour, giving the surgeon better procedural control and reducing procedure time(8). In 2015, Simona Mazzoni et al. further developed the computer-aided designing and manufacturing technique in fabricating surgical cutting guides and titanium fixation plates in upper maxilla repositioning surgery without an occlusal wafer. The study result confirmed the high accuracy in transferring the virtual planning by using the surgical guides and fixation plates(9).

In reviewing the literature, the application of 3D printing of titanium fixation plates in jaw surgery are available only at two centers currently: the Maxillofacial Surgery Department of S Orsola Malpighi Hospital in Italy and the Oral and Maxillofacial Surgery Department of Lund University in Sweden(6,7). The published preliminary work have proved the prospect of 3D-printed titanium plates in promoting mandibular reconstruction surgery and upper maxilla orthognathic surgery though their printed titanium plates looked rather bulky and the sample sizes were small and there is still lack of qualified randomized controlled trials between the printed and the conventional titanium plates. To better benefit from the burgeoning use of 3D printing in health care, we will develop a new designing and manufacturing protocol in printing customized fixation plates, which will be designed in specific loading circumstances and will perfectly adapt to the anatomical structures of the jaw. It is imperative to conduct a feasibility study in exploring the application of 3D printing of titanium fixation plates in jaw surgery based on our patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 of either gender; and
2. Signed informed consent form;and
3. Single or double-jaw orthognathic surgery under general anaesthesia, or
4. Jaw reconstruction due to benign or malignant tumor, osteomyelitis, and osteonecrosis under general anaesthesia.

Exclusion Criteria:

1. Unstable or complicated systemic diseases that contraindicate the surgical process.
2. Severe systemic diseases or conditions that would potentially compromise the healing process.
3. Patients who are pregnant.
4. Patients who are unable to take CT/CBCT scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Intraoperative success rate | Intraoperation
  1) the uneventful application of the 3D-printed patient-specific titanium plate in jaw surgery without any minor revision; 2) the final restored outcome being optimal based on clinical parameters.

SECONDARY OUTCOMES:
Incidence of postoperative adverse events [safety] | 2-5 years postoperation
  An adverse event is defined as any untoward medical occurrence in a patient administered the 3D-printed patient-specific titanium plate, which may or may not necessarily have a causal relationship with this new device.

OTHER OUTCOMES:
Accuracy | One and six months after surgery.
  The accuracy of using the 3D-printed customized titanium plates in transferring the virtual surgical plan.

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiong SU, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- The Prince Philip Dental Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martola M, Lindqvist C, Hanninen H, Al-Sukhun J. Fracture of titanium plates used for mandibular reconstruction following ablative tumor surgery. J Biomed Mater Res B Appl Biomater. 2007 Feb;80(2):345-52. doi: 10.1002/jbm.b.30603. PMID 16850467
- [Background] Sing SL, An J, Yeong WY, Wiria FE. Laser and electron-beam powder-bed additive manufacturing of metallic implants: A review on processes, materials and designs. J Orthop Res. 2016 Mar;34(3):369-85. doi: 10.1002/jor.23075. Epub 2015 Oct 29. PMID 26488900
- [Background] Parthasarathy J. 3D modeling, custom implants and its future perspectives in craniofacial surgery. Ann Maxillofac Surg. 2014 Jan;4(1):9-18. doi: 10.4103/2231-0746.133065. PMID 24987592
- [Background] Ventola CL. Medical Applications for 3D Printing: Current and Projected Uses. P T. 2014 Oct;39(10):704-11. PMID 25336867
- [Background] Derand P, Rannar LE, Hirsch JM. Imaging, virtual planning, design, and production of patient-specific implants and clinical validation in craniomaxillofacial surgery. Craniomaxillofac Trauma Reconstr. 2012 Sep;5(3):137-44. doi: 10.1055/s-0032-1313357. PMID 23997858
- [Background] Ciocca L, Mazzoni S, Fantini M, Persiani F, Marchetti C, Scotti R. CAD/CAM guided secondary mandibular reconstruction of a discontinuity defect after ablative cancer surgery. J Craniomaxillofac Surg. 2012 Dec;40(8):e511-5. doi: 10.1016/j.jcms.2012.03.015. Epub 2012 Apr 30. PMID 22551671
- [Background] Mazzoni S, Marchetti C, Sgarzani R, Cipriani R, Scotti R, Ciocca L. Prosthetically guided maxillofacial surgery: evaluation of the accuracy of a surgical guide and custom-made bone plate in oncology patients after mandibular reconstruction. Plast Reconstr Surg. 2013 Jun;131(6):1376-1385. doi: 10.1097/PRS.0b013e31828bd6b0. PMID 23714798
- [Background] Mazzoni S, Bianchi A, Schiariti G, Badiali G, Marchetti C. Computer-aided design and computer-aided manufacturing cutting guides and customized titanium plates are useful in upper maxilla waferless repositioning. J Oral Maxillofac Surg. 2015 Apr;73(4):701-7. doi: 10.1016/j.joms.2014.10.028. Epub 2014 Nov 29. PMID 25622881
- [Derived] Yang WF, Choi WS, Wong MC, Powcharoen W, Zhu WY, Tsoi JK, Chow M, Kwok KW, Su YX. Three-Dimensionally Printed Patient-Specific Surgical Plates Increase Accuracy of Oncologic Head and Neck Reconstruction Versus Conventional Surgical Plates: A Comparative Study. Ann Surg Oncol. 2021 Jan;28(1):363-375. doi: 10.1245/s10434-020-08732-y. Epub 2020 Jun 22. PMID 32572853
- [Derived] Yang WF, Choi WS, Zhu WY, Su YX. "One-piece" patient-specific reconstruction plate for double-barrel fibula-based mandibular reconstruction. Int J Oral Maxillofac Surg. 2020 Aug;49(8):1016-1019. doi: 10.1016/j.ijom.2019.12.006. Epub 2019 Dec 28. PMID 31892445
- [Derived] Yang WF, Zhang CY, Choi WS, Zhu WY, Li DTS, Chen XS, Du R, Su YX. A novel 'surgeon-dominated' approach to the design of 3D-printed patient-specific surgical plates in mandibular reconstruction: a proof-of-concept study. Int J Oral Maxillofac Surg. 2020 Jan;49(1):13-21. doi: 10.1016/j.ijom.2019.05.005. Epub 2019 Jun 21. PMID 31230767
- [Derived] Yang WF, Choi WS, Leung YY, Curtin JP, Du R, Zhang CY, Chen XS, Su YX. Three-dimensional printing of patient-specific surgical plates in head and neck reconstruction: A prospective pilot study. Oral Oncol. 2018 Mar;78:31-36. doi: 10.1016/j.oraloncology.2018.01.005. Epub 2018 Jan 16. PMID 29496055